CLINICAL TRIAL: NCT01879059
Title: The Effects of Altering Physical Activity on Endothelial Function, Glycemic Control, and the Blood Flow Response to an Oral Glucose Tolerance Test.
Brief Title: The Effects of Altering Physical Activity on Cardiometabolic Health
Acronym: PIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PIA-1200428
Record Dates: First submitted 2012-01-24; First posted 2013-06-17 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Insulin Resistance
Keywords: insulin resistance; exercise; continuous glucose monitoring; blood flow; endothelial function
MeSH Terms: conditions — Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): 5 days of inactivity followed by a 1 day return to physical activity
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — short period of inactivity (5 days) followed by a return to physical activity (1 day)

SUMMARY:
The effects of physical inactivity on variations in blood glucose and vascular health are not fully understood. The purpose of this study is to determine if an acute transition from physical activity to inactivity alters vascular health. Specifically, the investigators wish to examine in healthy, lean physically active individuals (obtaining greater than 10,000 steps/day) if decreasing physical activity (obtaining less than 5,000 steps/day) will alter blood flow following a meal a marker of vascular health. Furthermore, the investigators wish to examine if a one day return to physical activity (obtaining >10,000 steps/day) can restore the detrimental effects on blood flow following a meal.

DETAILED DESCRIPTION:
Herein, we tested the hypothesis that an acute reduction in daily activity (from >10,000 to <5,000 steps/day) for 5 days in healthy individuals reduced meal-stimulated blood flow and if a 1 day return to activity improved this outcomes.

ELIGIBILITY:
Inclusion Criteria:

* BMI: less than 30 kg/m2
* Physically active: exercise greater than 60mins per week

Exclusion Criteria:

* smoking
* type 2 diabetes
* Underlying conditions that limit ability to exercise safely
* Recent weight gain or loss(> 5% of body weight in 3 months)
* Recent (< 3 mo) changes in medication use or dose
* Pregnancy

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Thyfault, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Mikus CR, Oberlin DJ, Libla JL, Taylor AM, Booth FW, Thyfault JP. Lowering physical activity impairs glycemic control in healthy volunteers. Med Sci Sports Exerc. 2012 Feb;44(2):225-31. doi: 10.1249/MSS.0b013e31822ac0c0. PMID 21716152
- [Background] Mikus CR, Fairfax ST, Libla JL, Boyle LJ, Vianna LC, Oberlin DJ, Uptergrove GM, Deo SH, Kim A, Kanaley JA, Fadel PJ, Thyfault JP. Seven days of aerobic exercise training improves conduit artery blood flow following glucose ingestion in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Sep;111(3):657-64. doi: 10.1152/japplphysiol.00489.2011. Epub 2011 Jul 7. PMID 21737826

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: young, healthy, active men
Arm/Group | Exercise
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Effects of Physical Inactivity on Post Prandial Blood Flow
Description: There was a pre-measurement period of 3 days, then 5 days of inactivity, followed by 1.5-2 days of return to activity. A 10 day time frame overall. Blood flow measured by Doppler ultrasound during an oral glucose tolerance test before and after 5 days of inactivity.
Time Frame: 10 days
Population: healthy, young, active men
Measure: Mean (Standard Deviation); unit: percentage of change in blood flow
Arm/Group | Exercise
Number analyzed (Participants) | 13
percentage of change in blood flow | 0 (3)

ADVERSE EVENTS:
Arm/Group | Exercise
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No